CLINICAL TRIAL: NCT05136196
Title: Biomarker Stratified CaboZantinib (NSC#761968) and NivOlumab (NSC#748726) (BiCaZO) - A Phase II Study of Combining Cabozantinib and Nivolumab in Participants With Advanced Solid Tumors (IO Refractory Melanoma or HNSCC) Stratified by Tumor Biomarkers - an immunoMATCH Pilot Study
Brief Title: BiCaZO: A Study Combining Two Immunotherapies (Cabozantinib and Nivolumab) to Treat Patients With Advanced Melanoma or Squamous Cell Head and Neck Cancer, an immunoMATCH Pilot Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2021-12653; NCI-2021-12653 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S2101 (Other: SWOG); S2101 (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2021-11-25; First posted 2021-11-29 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-09

CONDITIONS: Clinical Stage III Cutaneous Melanoma AJCC v8; Clinical Stage III HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Clinical Stage IV Cutaneous Melanoma AJCC v8; Clinical Stage IV HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Locally Recurrent Head and Neck Squamous Cell Carcinoma; Locally Recurrent Hypopharyngeal Squamous Cell Carcinoma; Locally Recurrent Laryngeal Squamous Cell Carcinoma; Locally Recurrent Oral Cavity Squamous Cell Carcinoma; Locally Recurrent Oropharyngeal Squamous Cell Carcinoma; Metastatic Head and Neck Squamous Cell Carcinoma; Metastatic Hypopharyngeal Squamous Cell Carcinoma; Metastatic Laryngeal Squamous Cell Carcinoma; Metastatic Melanoma; Metastatic Oral Cavity Squamous Cell Carcinoma; Metastatic Oropharyngeal Squamous Cell Carcinoma; Recurrent Melanoma; Stage III Hypopharyngeal Carcinoma AJCC v8; Stage III Laryngeal Cancer AJCC v8; Stage III Lip and Oral Cavity Cancer AJCC v8; Stage III Oropharyngeal (p16-Negative) Carcinoma AJCC v8; Stage IV Hypopharyngeal Carcinoma AJCC v8; Stage IV Laryngeal Cancer AJCC v8; Stage IV Lip and Oral Cavity Cancer AJCC v8; Stage IV Oropharyngeal (p16-Negative) Carcinoma AJCC v8; Unresectable Melanoma
MeSH Terms: conditions — Oropharyngeal Neoplasms; Squamous Cell Carcinoma of Head and Neck; Melanoma; Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Mouth Neoplasms; Carcinoma | interventions — Biopsy; Specimen Handling; cabozantinib; Magnetic Resonance Spectroscopy; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (nivolumab and cabozantinib) (Experimental): Patients receive nivolumab IV over 30 minutes on day 1 of each cycle and cabozantinib PO daily. Cycles repeat every 28 days for 2 years in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or MRI scans and collection of blood samples throughout the trial. Patients undergo a tumor biopsy during screening and optionally during follow-up.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Drug: Cabozantinib S-malate; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo tumor biopsies
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Cabozantinib S-malate — Given PO
  Other Names: BMS-907351; Cabometyx; Cometriq; XL 184; XL-184; XL184
Procedure: Computed Tomography — Undergo CT scans
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI scans
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo

SUMMARY:
This phase II trial studies the good and bad effects of the combination of drugs called cabozantinib and nivolumab in treating patients with melanoma or squamous cell head and neck cancer that may have spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body (advanced). Cabozantinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. This trial may help doctors determine how quickly patients can be divided into groups based on biomarkers in their tumors. A biomarker is a biological molecule found in the blood, other body fluids, or in tissues that is a sign of a normal or abnormal process or a sign of a condition or disease. A biomarker may be used to see how well the body responds to a treatment for a disease or condition. The two biomarkers that this trial is studying are "tumor mutational burden" and "tumor inflammation signature." Another purpose of this trial is to help doctors learn if cabozantinib and nivolumab shrink or stabilize the cancer, and whether patients respond differently to the combination depending on the status of the biomarkers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the feasibility of molecular characterization based on tumor mutation burden (TMB) for participant stratification, as assessed by the proportion of participants with less than or equal to a 21-day turnaround time for biopsy results in Stage I of the study.

II. To evaluate the feasibility of molecular characterization based on TMB and gene expression profiling (GEP) (for Tumor Inflammation Score [TIS]) for stratification, as assessed by the proportion of participants with less than or equal to a 21-day turnaround time for biopsy results in Stage II of the study.

III. To evaluate the efficacy by overall response rate (ORR - defined as confirmed and unconfirmed partial responses plus complete responses) of cabozantinib S-malate (cabozantinib) plus nivolumab in each disease cohort, both across and within tumor biomarker subgroups.

SECONDARY OBJECTIVES:

I. To assess the difference in ORR in each disease cohort between tumor marker subgroups separately for each disease cohort.

II. To assess safety and tolerability of this treatment in these populations. III. To estimate disease control rate (DCR) in participants receiving cabozantinib plus nivolumab in each disease cohort, stratified by tumor biomarkers.

IV. To estimate progression-free survival (PFS) in participants receiving cabozantinib plus nivolumab in each disease cohort, stratified by tumor biomarkers.

V. To estimate overall survival (OS) in participants receiving cabozantinib plus nivolumab in each disease cohort, stratified by tumor biomarkers.

VI. To assess the proportion of patients with assay failure, and the time from the date of tissue collection to molecular group determination at the end of Stage I.

ADDITIONAL OBJECTIVE:

I. To identify candidate biomarkers predictive of response and toxicity to the cabozantinib and nivolumab combination.

BANKING OBJECTIVE:

I. To bank specimens for future correlative studies.

OUTLINE:

Patients receive nivolumab intravenously (IV) over 30 minutes on day 1 of each cycle and cabozantinib orally (PO) daily. Cycles repeat every 28 days for 2 years in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT) or magnetic resonance imaging (MRI) scans and collection of blood samples throughout the trial. Patients undergo a tumor biopsy during screening and optionally during follow-up.

After completion of study treatment, patients are followed up every 12 weeks for 1 year and then every 6 months until 3 years after step 2 registration.

ELIGIBILITY:
Inclusion Criteria:

* STEP 1 - SPECIMEN SUBMISSION
* Participants must have histologically confirmed melanoma that is stage III or IV, unresectable, recurrent, or metastatic non-uveal melanoma OR Participants must have histologically confirmed squamous cell carcinoma of the head and neck (HNSCC) that is either locally recurrent and non-amendable to curative therapy (e.g., radiation, surgery) or metastatic. The primary tumor location must be the oropharynx, oral cavity, hypopharynx, or larynx. Primary tumor site of nasopharynx (any histology) or unknown primary tumor are not eligible

  * Note: For participants with primary oropharyngeal cancer, human papillomavirus (HPV) or p16 status must be known prior to step 1 registration
* Participants must have disease presentation consistent with measurable disease. Note: Current disease measurements will not be required until step 2 registration
* Participants must have had documented progression during or within 12 weeks after the last dose of PD-1 checkpoint inhibition-based therapy. Participants must have been receiving checkpoint inhibition for a minimum of 6 weeks. Participants who recur during adjuvant anti-PD1 treatment or within 12 weeks of completion of adjuvant anti-PD1 treatment are eligible if they have measurable disease and are considered unresectable
* Participants with known human immunodeficiency virus (HIV)-infection must be receiving anti-retroviral therapy and have an undetectable viral load test within 6 months prior to step 1 registration
* Participants with evidence of chronic hepatitis B virus (HBV) infection must have undetectable HBV viral load within 28 days prior to step 1 registration
* Participants with a history of hepatitis C virus (HCV) infection must have no detectable viral load within 28 days prior to step 1 registration
* Participants must not have an active infection requiring systemic therapy (except HBV, HCV or HIV as mentioned above)
* Participants must not have experienced myocardial infarction or thromboembolic event requiring anticoagulation within 90 days prior to step 1 registration, unless clinically stable with ongoing medical management
* Participants must have recovered to baseline or =< grade 1 Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5 toxicities related to any prior treatments, unless adverse events are deemed clinically nonsignificant by the treating investigator or stable on supportive therapy
* Participants must not have received more than one prior primary radiotherapy regimen, curative or adjuvant, to the mucosal surfaces of the head and neck, with the additional following criteria:

  * If the primary radiation is combined with chemotherapy, a minimum of 16 weeks will be required to have elapsed between the end of radiotherapy and step 1 registration. If the radiation is given alone, a minimum of 8 weeks will be required to have elapsed between the end of radiotherapy and step 1 registration
  * Additional palliative radiotherapy regimens are permitted but cannot have been administered to previously treated tissue (i.e., overlapping fields are excluded) with the exception of central nervous system (CNS) radiation and must be completed at least 4 weeks prior to step 1 registration
  * Treatment areas should be healed with no sequelae from radiation therapy (RT) that would predispose to fistula formation
* Participants must not have received prior treatment with anti-VEGF therapies for any reason
* Participants must be >= 18 years of age
* Participants must have a Zubrod Performance Status 0 or 1
* Participants must have adequate cardiac function. Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, must have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification and must be class 2B or better to be eligible for this trial
* Participants must not have any known significant organ disfunction that, in the opinion of the treating investigator, may impact suitability for receiving combination nivolumab/cabozantinib treatment
* Participants must be able to take oral medication without breaking, opening, crushing, dissolving or chewing capsules
* Participants must not have malabsorption syndrome
* Participants must not have active autoimmune disease requiring systemic steroids (equivalent of > 10mg of prednisone) or other immune suppression. Exceptions:

  * Type 1 diabetes mellitus
  * Endocrinopathy only requiring hormone replacement
  * Skin disorders (e.g., vitiligo, psoriasis, or alopecia) not requiring systemic treatment
  * Conditions not expected to recur in the absence of an external trigger
* Participants must not have received an organ allograft
* Participants must not have a history of hemoptysis (defined as >= 1/2 tsp of bright red blood per day) or tumor bleeding within 90 days prior to step 1 registration
* Participants must not have any of the following criteria due to the possibility of increased risk for tumor bleeding with cabozantinib therapy:

  * Prior carotid bleeding
  * Tumors that invade major vessels (e.g., the carotid) as shown unequivocally by imaging studies
  * Central (e.g., within 2 cm from the hilum) lung metastases that are cavitary as shown unequivocally by imaging studies
  * Any prior history of bleeding related to the current head and neck cancer
  * History of gross hemoptysis (bright red blood of 1/2 teaspoon or more per episode of coughing) within 3 months
* Participants must not require concomitant anticoagulation with coumarin agents (e.g., warfarin), direct thrombin inhibitors (e.g., dabigatran), direct factor Xa inhibitor betrixaban, or platelet inhibitors (e.g., clopidogrel)

  * Participants must not require anticoagulants except for the following:

    * Prophylactic use of low-dose aspirin for cardio-protection (per local applicable guidelines) and low-dose low molecular weight heparins (LMWH).
    * Therapeutic doses of LMWH or anticoagulation with direct factor Xa inhibitors, rivaroxaban, edoxaban, or apixaban in participants without known brain metastases who are on a stable dose of the anticoagulant for at least 1 week prior to step 1 registration without clinically significant hemorrhagic complications from the anticoagulation regimen or the tumor
* Participants must not have evidence of preexisting uncontrolled hypertension 28 days prior to step 1 registration as documented by baseline blood pressure reading with systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 90 mmHg. Participants on antihypertensive therapies with controlled blood pressure are eligible
* Participants must not have a prior or concurrent malignancy whose natural history or treatment (in the opinion of the treating physician) has the potential to interfere with the safety or efficacy assessment of the investigational regimen
* Participants must not be pregnant or nursing due to the known safety profiles of the drugs in this study. Individuals who are of reproductive potential must have agreed to use an effective contraceptive method with details provided as a part of the consent process. A person who has had menses at any time in the preceding 12 consecutive months or who has semen likely to contain sperm is considered to be of "reproductive potential". In addition to routine contraceptive methods, "effective contraception" also includes refraining from sexual activity that might result in pregnancy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) including hysterectomy, bilateral oophorectomy, bilateral tubal ligation/occlusion and vasectomy with testing showing no sperm in the semen
* Have an adequate archival tissue specimen verified by the local pathologist and documented on the Pathology Review Form from a procedure obtained after the development of resistance to anti-PD-1/L1 therapy. Archival tissue must consist of tumor block or at least 1 hematoxylin and eosin (H&E)-stained 4-5 micron slide and 20 freshly cut serially sectioned and numbered 4-5 micron unstained, uncharged slides OR

Be willing to undergo research biopsy AND have tumor accessible for biopsy based on the following criteria:

* Mediastinal, laparoscopic, gastrointestinal, or bronchial endoscopic biopsies can be obtained incidentally to a clinically necessary procedure and NOT for the sole purpose of the clinical trial
* Acceptable biopsy procedures are:

  * Percutaneous biopsy with local anesthetic and/or sedation with an expected risk of severe complications < 2%
  * Direct transoral biopsy (with or without local anesthetic and/or sedation) with an expected risk of severe complications < 2%
  * Excisional cutaneous biopsy with local anesthetic and/or sedation with an expected risk of severe complications < 2%
  * Biopsy with removal of additional tumor tissue during a medically necessary mediastinoscopy, laparoscopy, gastrointestinal endoscopy, bronchoscopy or craniotomy. No open surgical, laparoscopic or endoscopic procedure should be performed solely to obtain a biopsy for this protocol
  * Removal of additional tumor tissue during a medically necessary surgical procedure

    * Participants must submit whole blood for germline genomic analysis
    * Participants must have been offered the opportunity to participate in specimen banking
    * Note: As a part of the Oncology Patient Enrollment Network (OPEN) registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system
* Participants must be informed of the investigational nature of this study and must sign and give informed consent in accordance with institutional and federal guidelines
* Participants with impaired decision-making capacity are eligible as long as their neurological or psychological condition does not preclude their safe participation in the study (e.g., tracking pill consumption and reporting adverse events to the investigator)

  * STEP 2 TREATMENT REGISTRATION
* Note: No tests or exams are required to be repeated for step 2 registration (Treatment). However, participants who are known to have a change in eligibility status after step 1 registration are not eligible for step 2 registration

  * Participants must continue to meet eligibility for step 1 registration prior to step 2 registration
  * Participants must have had their tumor tissue submitted via the Southwest Oncology Group (SWOG) Specimen Tracking System prior to step 2 registration
  * Participants registered during stage II of the protocol must have received assignment to an open cohort from the SWOG Statistics and Data Management Center based on their biomarker screening profile (not applicable for patients registered during stage I of the protocol)
  * Participants must have measurable disease. All measurable disease must be assessed within 28 days prior to step 2 registration. All non-measurable disease must be assessed within 42 days prior to step 2 registration. Note: All disease must be assessed and documented on the Baseline Tumor Assessment Form (Response Evaluation Criteria in Solid Tumors [RECIST] 1.1)
  * For melanoma participants, CT chest, abdomen and pelvis must be obtained. For HNSCC participants, CT neck and chest must be obtained. Further imaging (i.e., MR brain, CT abdomen/pelvis or extremities, bone scan) will be performed as deemed appropriate by the treating physician
  * Participants with treated brain metastases must have no evidence of progression on the follow-up brain imaging after central nervous system (CNS)-directed therapy
  * Participants must not have experienced any significant health changes that, in the opinion of the treating investigator, may impact continued suitability for receiving combination nivolumab/cabozantinib treatment
  * Participants with treated brain metastases must have discontinued steroid treatment at least 14 days prior to step 2 registration
  * Participants must not have received investigational agents or monoclonal antibodies (except Food and Drug Administration [FDA] approved supportive care antibodies, such as denosumab) within 28 days prior to step 2 registration
  * Participants must not have received surgery, chemotherapy, radiation therapy, biologic agents, or steroids within 14 days prior to step 2 registration
  * Participants must not have received administration of a live, attenuated vaccine within 30 days prior to step 2 registration. Note: Participants may have received a messenger ribonucleic acid (mRNA) or viral vector-based coronavirus disease 2019 (COVID-19) vaccine within 30 days prior to step 2 registration
  * Participants must not have received administration of any strong CYP3A4 inducers, such as but not limited to rifampin, carbamazepine, enzalutamide, mitotane, phenytoin and St. John's wort, within 14 days prior to step 2 registration
  * Participants must not have received administration of any strong CYP3A4 inhibitors, such as but not limited to clarithromycin, itraconazole, ketoconazole, grapefruit juice, indinavir, nelfinavir, ritonavir, nefazodone, saquinavir, and telithromycin, within 5 times the half-life of the CYP3A inhibitor prior to step 2 registration
  * Participants must have a history and physical examination performed within 28 days prior to step 2 registration
  * Leukocytes >= 3,000/uL (within 28 days prior to step 2 registration)
  * Absolute neutrophil count >= 1,500/uL (within 28 days prior to step 2 registration)
  * Platelets >= 100,000/uL (within 28 days prior to step 2 registration)
  * Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) or =< 3 x ULN for participants with Gilbert's disease (within 28 days prior to step 2 registration)
  * Aspartate aminotransferase (AST) =< 3 x institutional ULN (within 28 days prior to step 2 registration)
  * Alanine aminotransferase (ALT) =< 3 x institutional ULN (within 28 days prior to step 2 registration)
  * Urinalysis: For baseline value (no required value for eligibility)
  * Measured (OR calculated) creatinine clearance >= 30 mL/min using the following Cockcroft-Gault Formula. This specimen must have been drawn and processed within 28 days prior to step 2 registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-12-06 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Biomarker results turnaround time | Within 21 days
  A biomarker turnaround time estimate of at least 75% within 21 days will be considered successful with respect to feasibility. For melanoma participants, turnaround time is defined as the time-period between date of tissue submission by the site to central repository and date the site was sent notification of participant molecular group determination. For head and neck squamous cell carcinoma (HNSCC) participants, turnaround time is defined as the time-period between date of tissue submission by the site to central repository and one day after both results have been received by the Southwest Oncology Group Statistics and Data Management Center to simulate when the site would have received notification of participant molecular group determination.
Objective response rate | At the end of stage I
  Confirmed and unconfirmed complete and partial responses) in molecular subgroups. Will assess biomarker response association. To test this association, will consider combination of biomarkers coded as 0 = Lo/Lo, 1 = Lo/Hi or Hi/Lo, and 2 = Hi/Hi. Assume each biomarker level is associated with an odds-ratio of approximately 3.1 (for example, corresponding to a difference in response rate of 5 percent to 14 percent from Lo/Lo to Lo/Hi or Hi/Lo). For the melanoma cohort, with approximately equal sized biomarker combination subgroups, a one-sided 0.10 level test for trend using (0,1,2) coding with logistic regression has a power of 80%. The same analysis for HNSCC will have lower power for the same effect size due to the unequal frequencies in the subgroups defined by the biomarkers. We will also conduct disease-by-biomarker interaction tests; however, there will be limited power to detect even to detect relatively large interaction parameters.

SECONDARY OUTCOMES:
Rate and profile of >= grade 3 treatment-related adverse events | Up to 2 years
  Per Common Terminology Criteria for Adverse Events 5.0. With respect to overall disease group, 60 participants are sufficient to estimate the probability of a particular toxicity to within +/- 13 percent. Any toxicity occurring with at least a 5 percent probability is likely to be seen at least once (95 percent chance).
Disease control rate | Up to 2 years
  Will be estimated using the method of Kaplan-Meier.
Progression-free survival | From date of registration to date of first documentation of progression or symptomatic deterioration, or death due to any cause, assessed up to 2 years
  Will be estimated using the method of Kaplan-Meier.
Overall survival | From date of registration to date of death due to any cause, assessed up to 2 years
  Will be estimated using the method of Kaplan-Meier.
Turnaround time for the Tumor Inflammation Score in stage II | Assessed within 21 days

OTHER OUTCOMES:
Additional markers of response or resistance | Up to 2 years
  Explore additional markers of response or resistance through hypothesis generating analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Siwen Hu-Lieskovan, Principal Investigator — SWOG Cancer Research Network
Locations (213):
- United States (213):
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Tower Cancer Research Foundation, Beverly Hills, California
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - The Angeles Clinic and Research Institute - West Los Angeles Office, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Rocky Mountain Regional VA Medical Center, Aurora, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Cancer Care and Hematology-Fort Collins, Fort Collins, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Rush-Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Memorial Hospital East, Shiloh, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - Tufts Medical Center, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo Cancer Center, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Saint Mary's - Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Essentia Health - Fosston, Fosston, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Essentia Health - Park Rapids, Park Rapids, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Essentia Health - Jamestown Clinic, Jamestown, North Dakota
  - Miami Valley Hospital South, Centerville, Ohio
  - Premier Blood and Cancer Center, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Miami Valley Cancer Care and Infusion, Greenville, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Jefferson Torresdale Hospital, Philadelphia, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Dartmouth Cancer Center - North, Saint Johnsbury, Vermont
  - Inova Alexandria Hospital, Alexandria, Virginia
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Inova Fair Oaks Hospital, Fairfax, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Centra Alan B Pearson Regional Cancer Center, Lynchburg, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - VCU Health Tappahannock Hospital, Tappahannock, Virginia
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Essentia Health Saint Mary's Hospital - Superior, Superior, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm